CLINICAL TRIAL: NCT02535520
Title: Clinical Evaluation of RTVue XR With SSADA in Retinal Patients
Brief Title: Evaluation of RTVue XR With SSADA
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Sponsor
Other Study IDs: 200-50547
Record Dates: First submitted 2015-08-26; First posted 2015-08-28 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2015-10

CONDITIONS: Retina Vascular Pathology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Optovue has implemented a motion contrast imaging software in RTVue XR, a split spectrum amplitude decorrelation algorithm (SSADA), for non-invasive imaging of ocular vasculature. Consented subjects will undergo a series of images of the back of the eye using an Optical Coherence Tomograpy (OCT) device, RTVue XR, in addition to the conventional images as part of clinical routine. SSADA images will be compared with conventional methods.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Able and willing to complete exams
* Patients in retina clinic that need angiography

Exclusion Criteria:

* Unable to complete the required examinations and visits
* Large amount of subretinal hemorrhage
* Media opacity leading to poor quality images
* Extreme refractive error leading to poor quality images
* Pathologies in the anterior segment leading to poor quality images

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seeing eye doctor for routine or follow-up care
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Agreement of SSADA to conventional angiography | Day 1